CLINICAL TRIAL: NCT05795218
Title: A Prospective, Multi-center, Single Arm, Observational, Post-market Clinical Follow-up Study on the Use of the directSTIM™ Deep Brain Stimulation System to Treat Essential Tremor
Brief Title: directSTIM™ Deep Brain Stimulation System Post-Market Clinical Follow-up Study on Essential Tremor
Status: Terminated | Type: Observational
Why Stopped: Insolvency of the business
Sponsor: Aleva Neurotherapeutics SA (Industry)
Responsible Party: Sponsor
Other Study IDs: CLI-12082
Record Dates: First submitted 2022-07-05; First posted 2023-04-03 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2023-07

CONDITIONS: Essential Tremor
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Essential Tremor | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Deep Brain Stimulation — implant and DBS therapy with the directSTIM™ DBS system
  Other Names: DBS

SUMMARY:
This is a prospective, multi-center, single arm post-market clinical follow-up study.

The present study investigates a product authorized on the European market that will be used per its intended use, and all procedures involved follow the standard of care.

This is an observational study to provide clinical evidence in support of DBS effectiveness in the treatment of ET when delivered by the directSTIM DBS system.

Twenty-one patients will be enrolled in this study. Subjects selected to participate in the study will be ET patients referred to uni- or bilateral DBS implant who meet the inclusion criteria and none of the exclusion criteria.

Primary effectiveness variables will be measured at baseline for the identification of the worst limb (most affected by the disease), then 3 months post-surgery. Safety events will be collected between implant and 3-month visit, to evaluate potential confounding factors.

After completing the 3-month visit, subjects will exit the study, and continue to be followed by their physician per usual care.

Study will be conducted at minimum 3 centers in Europe.

DETAILED DESCRIPTION:
This study investigates the benefits and safety of the use of the directSTIM Deep Brain Stimulation (DBS) system within its intended use, to deliver DBS therapy to patients suffering from Essential Tremor (ET) whose motor symptoms are no longer optimally controlled through pharmaceutical treatment.

The objective of this study is to show that directSTIM is not inferior to competitor DBS Systems at alleviating postural or kinetic symptoms of Essential Tremor through the delivery of Deep Brain Stimulation therapy.

Data to be analyzed will be collected from ET patients referred for DBS surgery, who chose to get the directSTIM DBS System implanted after discussing its risks and benefits with their clinician.

All procedures involving the patient and the device follow the standard of care in place at the site for DBS.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older.
* Patient with main tremor symptoms in upper limbs.
* Patient was referred for DBS surgery to treat Essential Tremor and chose the directSTIM DBS System
* Patient has a postural or kinetic tremor severity score of at least 3 out of 4 in the extremity intended for treatment on the Fahn-Tolosa-Marin Clinical Rating Scale for Tremor with medication, for the worst limb (i.e. most affected by disease)
* Patient accepts to abstain from caffeine for 8 hours and from alcohol for 12 hours before visit.
* Patient accepts to turn stimulation off for 1 hour prior to the 3-month follow-up visit.
* Patient is willing to provide a written informed consent.
* Patient is available for the study visit, and other study requirements.

Exclusion Criteria:

* Cognitive impairment, or any characteristic that would limit study candidate's ability to complete study assessments, such as:

  * Active major psychiatric disorder (including clinically significant depression as rated by the clinician)
  * Patient had dementia interfering with their ability to co-operate or comply with study requirements or comprehend the informed consent (mini-mental exam score <24 or otherwise not capable of discernment)
  * Presence of an electrical or electromagnetic implant (e.g. cochlear implant, pacemaker)
  * Previous brain ablation/surgical procedure
  * Neurological injury, evidence of supraspinal central nervous system disease
  * History of seizures
  * Diathermy
  * Abuse of drugs or alcohol.
* Patient had botulinum toxin injection less than 6 months prior to enrollment
* Patient is participating in another clinical study that would confound data analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty-one patients suffering from Essential Tremor, referred for DBS surgery, who chose directSTIM, will be enrolled in a minimum of 3 sites in Europe to collect primary safety and effectiveness variables baseline and 3 months post-surgery.
  The sample size has been determined for the primary effectiveness endpoint. Study subjects will be representative of the target population since they will be recruited among patients who discussed the need and agreed with their clinician upon the implant of a DBS System to treat their motor symptoms caused by Essential Tremor.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Change in the motor performance subscale of the Fahn Tolosa Marin Essential Tremor Rating Scale (FTM ETRS) score of target limb | 3 months
  The motor scale of the Fahn Tolosa Marin Essential Tremor Rating Scale (FTM ETRS) measures the maximum tremor severity in various body regions in different positions (rest, postural, kinetic).
  Each body area is evaluated in Part A of the FTM ETRS, which is composed of 10 questions.
  The FTM ETRS utilizes a 0 to 4 point scale where 0 indicates non-symptomatic (normal) and 4 indicates the most severe rating of the patient's tremor symptoms.
  The target limb (arm) will be identified at baseline for each patient as the limb most severely affected by tremors (highest score in postural or kinetic assessment in part A).
  The primary efficacy outcome is the mean percentage difference, 3 months post-implant, between the with and without stimulation states, as measured on the target limb identified at baseline, by the individual performance subscale score (i.e. postural or kinetic) on the FTM ETRS.

SECONDARY OUTCOMES:
Proportions of Adverse Events and Device Deficiencies observed | 3 months
  Proportions of the following events from DBS implant through study completion:
  * Adverse Events:
    * Surgery-related
    * Device-related
    * Therapy-related
  * Device deficiencies
Change in total motor score on the Fahn Tolosa Marin Essential Tremor Rating Scale | 3 months
  The motor scale of the Fahn Tolosa Marin Essential Tremor Rating Scale (FTM ETRS) measures the maximum tremor severity in various body regions in different positions (rest, postural, kinetic).
  FTM ETRS is divided into 3 parts (A, B and C). The total motor score is calculated by summation of the individual scores to questions 1-15 of parts A and B.
  Maximum score of Part A is 88 points while that of Part B is of 36 points.
  The secondary efficacy OBJECTIVE is the mean difference between the with and without stimulation states, 3 months post-implant, as measured by the total motor score on the FTM ETRS.
  A high total motor score (i.e. close to 124) indicates overall poor motor performance - i.e. severe tremor.
  High difference value between total motor score measured with and without stimulation indicates a strong improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Michalis, Study Director — Aleva Neurotherapeutics SA
Locations (5):
- Germany (5):
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Münster, Münster

IPD SHARING:
Plan to Share IPD: No